CLINICAL TRIAL: NCT01159028
Title: A Phase I Clinical Trial to Study the Safety, Pharmacokinetics, and Efficacy of BP1001 (L-Grb-2 Antisense Oligonucleotide) in Patients With Refractory or Relapsed Acute Myeloid Leukemia, Philadelphia Chromosome Positive Chronic Myelogenous Leukemia, or Acute Lymphoblastic Leukemia, and Myelodysplastic Syndrome
Brief Title: Clinical Trial of BP1001 (L-Grb-2 Antisense Oligonucleotide) in CML, AML, ALL & MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Path Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0578 (v) 08-8
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome; Ph1 Positive CML
Keywords: Liposomal Grb-2 treatment of CML, AML, CLL, MDS; Liposomal Grb-2 with LDAC for AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BP1001 (Experimental): Subjects are treated with open-label study drug (BP1001) in a dose-escalation model.
  Interventions: Drug: BP1001
- BP1001 in combination with LDAC (Experimental): AML subjects are treated with open-label escalating study drug (BP1001) in combination with low dose ara-C (LDAC)
  Interventions: Drug: BP1001 in combination with LDAC

INTERVENTIONS:
Drug: BP1001 — Study drug (BP1001) is constituted in normal saline, administered by IV on twice weekly for 28 days.
  Other Names: Liposomal Grb-2; L-Grb-2; BP-100-1.01
  Arms: BP1001
Drug: BP1001 in combination with LDAC — Study drug (BP1001) is constituted in normal saline, administered by IV twice weekly for 28 days. Low dose ara-C (LDAC) is self administered twice daily for 10 consecutive days during the 28 day cycle.
  Other Names: Liposomal Grb-2; L-Grb-2; BP-100-1.01; low dose ara-C
  Arms: BP1001 in combination with LDAC

SUMMARY:
The first goal of this clinical research study is to find the highest safe dose of BP1001, a liposomal Growth Factor Receptor Bound Protein-2 antisense oligodeoxynucleotide (L-Grb2 AS), for patients with Philadelphia Chromosome positive CML, AML, ALL and MDS. The response of the leukemia to this treatment will also be studied. The second goal of this clinical research study is to evaluate the safety and toxicity of the combination of BP1001 and concurrent low-dose ara-C (LDAC) in patients with AML.

DETAILED DESCRIPTION:
The Philadelphia Chromosome is an unusual genetic trait found in 90-95% of patients with CML and approximately 20-25% of patients with ALL. The protein created by this unusual trait causes normal cells within the body to become cancer cells, and then causes these cells to grow and divide at a rapid rate. Researchers think that the protein "Growth Factor Receptor Bound Protein-2 (Grb-2)" plays an important role in the rapid growth of leukemic cells. The study drug (BP1001) may be able to inhibit the cells from making Grb-2. Researchers hope that without this protein, the leukemia cells will die.

Up to 60 patients are expected to be enrolled on this study.

Part A: Dose escalation: Each cohort will receive BP1001 at a dose higher than the previous group.

Part B: Dose-expansion Cohorts: Subjects with relapsed or refractory AML will receive escalating doses of BP1001 concurrently with fixed low-dose ara-C (LDAC)

The study drug is an antisense molecule complementary to the messenger RNA (mRNA) code for the cell's expression of the protein Grb-2. The study drug is incorporated into lipid (fat) particles known as liposomes. This incorporation process is part of the manufacturing process and is done before the study drug is administered. The liposomes (which carry the study drug) will be administered intravenously twice a week for 28 days. Subjects enrolled in Part B of the study will receive study drug twice a week for 28 days concurrently with low dose ara-C, self administered twice daily for 10 consecutive days.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients 18 years of age or older
2. A diagnosis of refractory or relapsed AML, or Ph+ CML (in chronic, accelerated or blast phase, or acute lymphoblastic leukemia, or myelodysplastic syndrome.

   One of the following parameters is required to meet criteria for accelerated phase CML:
   * Blasts in Peripheral Blood or Bone Marrow ≥15%
   * Promyelocytes and Blasts in Peripheral Blood or Bone Marrow ≥30%
   * PB or BM basophils ≥20%
   * Thrombocytopenia <100 x 103/ml, not resulting from therapy

   Blast phase is defined as ≥30% blasts in peripheral blood or bone marrow, or presence of extramedullary disease, except for liver or spleen.
3. Patients with CML must have demonstrated resistance and/or intolerance to therapy with at least 2 tyrosine kinase inhibitors (TKI)
4. Patients with AML and ALL should have received at least 1 prior treatment regimen and either failed to achieve response or relapsed on treatment
5. Patients with MDS should have failed prior therapy with a hypomethylating agent or, if associated with a 5q- chromosomal abnormality, lenalidomide. NOTE: Patients with 5q- unable to receive or intolerant to lenalidomide are also eligible.
6. Have clinically adequate hepatic and renal functions as defined by:

   * ALT<2x ULN
   * Serum creatinine concentration <2x ULN
   * Serum bilirubin <2x ULN
7. Patients must sign an informed consent
8. Women of childbearing age must have a negative serum or urine pregnancy test prior to the initiation of study drug.
9. Barrier contraceptive precautions are to be used throughout the trial by all study participants of child bearing potential.
10. Have not received anti-cancer therapy for at least 2 weeks prior to study entry, with the exception of low dose ara-C (LDAC) given as subcutaneous injections (no less than 15 days prior), hydroxyurea or anagrelide (no less than 24 hours prior), TKI (no less than 5 days prior), and interferon (no less than 2 weeks prior)
11. Have an ECOG Performance of 0-2
12. Have a life-expectancy ≥3 months

Exclusion Criteria

1. Serious intercurrent medical illnesses which would interfere with the ability of the patient to carry out the treatment program
2. Pregnant or breastfeeding women
3. Patients who have uncontrolled active infection
4. Patients who have received another investigational product within the longer of 14 days or 5 half-lives of the previous product
5. Any history of adverse reaction or hypersensitivity to LDAC

Part B: BP1001 with Concurrent LDAC Dose-Expansion Cohorts

Enrollment in the dose-expansion cohorts (DEC) will be limited to only those patients with a diagnosis of refractory or relapsed AML(except acute promyelocytic leukemia) or those who are refractory to at least 1 prior therapy regimen and no more than 1 prior salvage regimen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Safety of BP1001 | 30 days
  Evaluate toxicity, tolerance, and MTD of escalating doses of BP1001
Safety of BP1001 in combination with LDAC | 30 days
  Evaluate safety and toxicity of the combination of BP1001 and concurrent LDAC using non-hematologic and hematologic measures per NCI CTCAE criteria.

SECONDARY OUTCOMES:
Optimal biologically active dose | 30 days
  Determine the optimal biologically active dose of BP1001 defined as a 50% reduction in Grb-2 expression in circulating leukemia cells
In vivo pharmacokinetics | 30 days
  Evaluate the in vivo PK of BP1001 in all subjects using plasma and urine to compute half life and elimination
Correlate PK data with historical experience | 30 days
  Correlate the in vivo PK data with historical experience to demonstrate the liposomal delivery performs as expected for all subjects by comparing PK data (half life and elimination) obtained from each subject with historical experience

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — M.D. Anderson Cancer Center; Maro Ohanian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Ohanian M, Tari Ashizawa A, Garcia-Manero G, Pemmaraju N, Kadia T, Jabbour E, Ravandi F, Borthakur G, Andreeff M, Konopleva M, Lim M, Pierce S, O'Brien S, Alvarado Y, Verstovsek S, Wierda W, Kantarjian H, Cortes J. Liposomal Grb2 antisense oligodeoxynucleotide (BP1001) in patients with refractory or relapsed haematological malignancies: a single-centre, open-label, dose-escalation, phase 1/1b trial. Lancet Haematol. 2018 Apr;5(4):e136-e146. doi: 10.1016/S2352-3026(18)30021-8. Epub 2018 Mar 14. PMID 29550383